CLINICAL TRIAL: NCT02450318
Title: Acute Vascular Response to Exercise in Women With Nonobstructive Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB201500077
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Nonobstructive Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Slow-paced walking (Experimental): Subjects will complete 47 minutes of walking at slow pace.
  Interventions: Other: Slow-paced walking

INTERVENTIONS:
Other: Slow-paced walking — Subjects will walk on a treadmill at a slow pace for 47 minutes

SUMMARY:
The purpose of this study is to examine the acute effect of exercise on vascular function in women with nonobstructive coronary artery disease.

DETAILED DESCRIPTION:
Women are more likely to have nonobstructive coronary artery disease (CAD) . The purpose of this study is to examine the acute effect of exercise on vascular function in women with nonobstructive coronary artery disease. Endothelium-dependent and -independent dilation, arterial stiffness and wave reflection will be measured at baseline and after walking on a treadmill at a slow pace for 47 minutes. Endothelium-dependent dilation will be measured using brachial artery flow-mediated dilation via high resolution ultrasonography. Endothelium-independent dilation will be measured using brachial artery dilation to sublingual nitroglycerin. Arterial stiffness and wave reflection will measured using applanation tonometry.

ELIGIBILITY:
Inclusion Criteria:

* women with non-obstructive coronary artery disease documented within the past 5 years by coronary angiogram as no coronary arteries with stenosis greater than 50% lesions
* age 18 to 89 years
* able to complete maximal graded exercise test

Exclusion Criteria:

* use of tobacco products within the previous six months
* use of oral contraceptives or hormone replacement therapy within the prior year
* pregnancy (positive urine pregnancy test) or lactation
* history of hepatic disease or infection with hepatitis B, C or HIV

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Change in endothelium-dependent dilation | Baseline, 15 minutes after exercise and 1 hour after exercise
  Brachial artery endothelium-dependent flow-mediated dilation to reactive hyperemia will be measured using high resolution ultrasonography. To determine flow-mediated dilation, brachial artery diameter and blood velocity will be measured before and after occluding the forearm for 5 minutes by inflating a cuff to 250 mmHg.

SECONDARY OUTCOMES:
Change in endothelium-independent dilation | Baseline, 15 minutes after exercise
  To determine vascular smooth muscle responsiveness to nitric oxide, brachial artery diameter will be measured using high resolution ultrasonography before and after sublingual administration of 0.4mg nitroglycerin.
Change in arterial stiffness and wave reflection | Baseline, 15 minutes after exercise and 1 hour after exercise
  Aortic pulse wave velocity and augmentation index will be measured using applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Demetra Christou, PhD, Principal Investigator — University of Florida
Locations (1):
- Integrative Cardiovasculal Physiology Laboratory, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No